CLINICAL TRIAL: NCT03692156
Title: Morphological Study of the Great Auricular Nerve and Adjacent Structures by Ultrasound Imaging and Transcutaneous Nerve Stimulation
Brief Title: Ultrasonic Morphological Study of the Great Auricular Nerve and Adjacent Structures
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xin Jiang, MD (Other)
Responsible Party: Sponsor-Investigator, Xin Jiang, MD, Principal Investigator, Shanghai Changzheng Hospital
Organization: Shanghai Changzheng Hospital (Other)
Other Study IDs: CHANGZHENG2018-15
Record Dates: First submitted 2018-09-27; First posted 2018-10-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-04

CONDITIONS: Great Auricular Nerve
Keywords: sternocleidomastoid muscle; Superficial Cervical Plexus block; ultrasound

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Ultrasound-guided nerve block has the characteristics of high success rate, few complications, and high patient satisfaction. It has been widely used in brachial plexus and lumbar plexus nerve blocks. Studies of ultrasound-guided superficial cervical plexus block are mostly unsatisfactory, and may be due to anatomic localization of the puncture site rather than real-time ultrasound guidance. The great auricular nerve is the largest branch of the superficial cervical plexus and may be identified under ultrasound. The aim of this study is to establish the success rate of identification of the great auricular nerve by combining ultrasound imaging with transcutaneous nerve stimulation. In addition, we will study the relationship between the success rate of identification and the related factors of patients. Another purpose of this study is to locate the position where the great auricular nerve emerges the posterior border of the sternocleidomastoid muscle. The relationship between this point and the midpoint of posterior border of the sternocleidomastoid muscle and adjacent structures will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing surgery in changzheng hospital

Exclusion Criteria:

* Suffering from malignant tumors, poor overall condition
* Communication barriers, unable to objectively describe symptoms
* Huge mass in the neck

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent surgery in our hospital during the study, especially neck surgery, such as cervical surgery, thyroid surgery, and carotid endarterectomy.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-03-30 (Estimated); Study Completion 2020-05-31 (Estimated)

PRIMARY OUTCOMES:
Success rate of identification of the great auricular nerve combining ultrasound imaging with transcutaneous nerve stimulation | 1 year
  Proportion of patients who's great auricular nerve was identified by combining ultrasound imaging with transcutaneous nerve stimulation

SECONDARY OUTCOMES:
Difference in gender | 1 year
  Patients were divided into two groups according to whether they recognized the great auricular nerve or not, and the differences in gender composition were compared.
Difference in BMI | 1 year
  Patients were divided into two groups according to whether they recognized the great auricular nerve or not, and the differences in BMI were compared.
Difference in body fat rate | 1 year
  Patients were divided into two groups according to whether they recognized the great auricular nerve or not, and the differences in body fat rate were compared.
Difference in neck circumference | 1 year
  Patients were divided into two groups according to whether they recognized the great auricular nerve or not, and the differences in neck circumference were compared.
Success rate of identification of the great auricular nerve by ultrasound | 1 year
  Proportion of patients who's great auricular nerve was identified by ultrasound
Distance between GAP and M | 1 year
  the distance between the point where the great auricular nerve emerges the posterior border of the sternocleidomastoid muscle and the midpoint of posterior border of the sternocleidomastoid muscle
SCM length | 1 year
  length of the posterior border of the sternocleidomastoid muscle

CONTACTS AND LOCATIONS:
Locations (1):
- Changzheng Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided